CLINICAL TRIAL: NCT05687357
Title: Tislelizumab in Combination With Pre-operative Chemoradiotherapy Versus SOC for Patients With Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma: a Multicenter, Randomized, Open-label, Phase IIB Trial
Brief Title: Tislelizumab in Combination With Pre-operative CRT Versus SOC for Locally Advanced G/GEJ Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-2010-IIT
Record Dates: First submitted 2022-12-26; First posted 2023-01-18 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2022-10

CONDITIONS: Gastric Cancer; Gastroesophageal-junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab; S 1 (combination); Oxaliplatin; Taxes; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Tislelizumab + Chemoradiotherapy (Experimental): Neoadjuvant: Prior to surgery, participants receive 4 cycles of Tislelizumab 200 mg via intravenous (IV) infusion on C1D1, C2D1, C2D22, C3D1 PLUS radiotherapy (TOMO or VMAT) 45Gy/1.5f PLUS S-1 initial dose depends on the body surface area, PO, bid, C1D1~D14，C2D1~C2D5, C2D8~C2D12, C2D15~C2D19, C2D22~C2D26, C2D29~C2D33, C3D1~D14 and oxaliplatin 130mg/m^2, IV, C1D1 and C3D1 OR S-1 initial dose depends on the body surface area, PO, bid, C1D1~D14，C3D1~D14 and nab-paclitaxel, IV 100~120mg/m^2，IV，C1D1，C1D8，C2D1，C2D8，C2D16，C2D22，C3D1 and C3D8.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive 3 cycles of SOX OR S-1 and nab-paclitaxel AND 3 cycles of S-1, AND up to 16 cycles of Tislelizumab 200 mg via IV infusion on Day 1 Q3W.
  Interventions: Drug: Tislelizumab; Drug: S-1; Drug: Oxaliplatin; Drug: Nab paclitaxel; Radiation: Radiation
- Arm B: Chemoradiotherapy (Active Comparator): Neoadjuvant: Prior to surgery, participants receive radiotherapy (TOMO or VMAT) 45Gy/1.5f PLUS S-1 initial dose depends on the body surface area, PO, bid, C1D1~D14，C2D1~C2D5, C2D8~C2D12, C2D15~C2D19, C2D22~C2D26, C2D29~C2D33, C3D1~D14 and oxaliplatin 130mg/m^2, IV, C1D1 and C3D1 OR S-1 initial dose depends on the body surface area, PO, bid, C1D1~D14，C3D1~D14 and nab-paclitaxel, IV 100~120mg/m^2，IV，C1D1，C1D8，C2D1，C2D8，C2D16，C2D22，C3D1 and C3D8.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive 3 cycles of SOX OR S-1 and nab-paclitaxel AND 3 cycles of S-1.
  Interventions: Drug: S-1; Drug: Oxaliplatin; Drug: Nab paclitaxel; Radiation: Radiation
- Arm C: Chemotherapy (Active Comparator): Neoadjuvant: S-1 initial dose depends on the body surface area, PO, bid, D1~D14，Q 3W for 6 cycles, and oxaliplatin 130mg/m^2, IV, D1 of each cycle for 6 cycles OR nab-paclitaxel, IV 100~120mg/m^2，IV，D1 and D8 for each cycle for 6 cycles.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive 3 cycles of SOX OR S-1 and nab-paclitaxel AND 3 cycles of S-1.
  Interventions: Drug: S-1; Drug: Oxaliplatin; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Tislelizumab — IV infusion
  Arms: Arm A: Tislelizumab + Chemoradiotherapy
Drug: S-1 — Oral tablets
Drug: Oxaliplatin — IV infusion
Drug: Nab paclitaxel — IV infusion
Radiation: Radiation — TOMO/VMAT
  Arms: Arm A: Tislelizumab + Chemoradiotherapy; Arm B: Chemoradiotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of Tislelizumab in the neoadjuvant (prior to surgery) or adjuvant (after surgery) treatment of previously untreated adults with gastric and gastroesophageal junction (GEJ) adenocarcinoma.

The primary study hypotheses are that:

Neoadjuvant and adjuvant Tislelizumab plus chemoradiotherapy, followed by adjuvant Tislelizumab and chemotherapy is superior to neoadjuvant chemoradiotherapy or chemotherapy, followed by adjuvant chemotherapy in terms of rate of Pathological Complete Response (pathCR) at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Has previously untreated localized gastric or GEJ adenocarcinoma as defined by T3~4aN+M0 or T4bNanyM0 （AJCC Version 8）
2. Has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1
3. Has adequate organ function.
4. Male participants of childbearing potential must agree to use an adequate method of contraception for the course of the study through 180 days after the last dose of chemotherapy.
5. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is greater.

Exclusion Criteria:

1. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that have undergone potentially curative therapy are not excluded.
2. Has received prior systemic anti-cancer therapy including investigational agents for the current malignancy.
3. Has an active infection requiring systemic therapy.
4. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
5. Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior the first dose of study treatment.
7. Has an active autoimmune disease that has required systemic treatment in past 2 years.
8. Has a known history of human immunodeficiency virus (HIV) infection.
9. Has a known history of Hepatitis B or known active Hepatitis C virus infection (HBsAg positive with HBV DNA≥500 IU/ml；HCV：HCV antigen positive with HCV copies >ULN).
10. Has had an allogenic tissue/solid organ transplant.
11. Has received a live vaccine within 30 days prior to the first dose of study treatment.
12. Female participants who are breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pathCR) Rate | Up to approximately 22 weeks
  PathCR rate is defined as the percentage of participants having a pathCR. pathCR is defined as no invasive disease within an entirely submitted and evaluated gross lesion, and histologically negative nodes.

SECONDARY OUTCOMES:
Event-free Survival (EFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 2 years
  EFS is based on RECIST 1.1 as assessed by the investigator and is defined as the time from randomization to the first of the following events: radiographic disease progression per RECIST 1.1; local or distant recurrence as assessed by CT scan or biopsy if indicated (for participants who are disease free after surgery); clinical progression as evidenced by peritoneal carcinomatosis confirmed by preoperative laparoscopy or laparotomy (for participants who are confirmed to be free of peritoneal involvement by laparoscopy at screening); or death due to any cause. A second primary malignancy, or radiographic progressive disease (PD) during the neoadjuvant phase that does not preclude successful surgery (i.e., disease free after surgery), are not considered EFS events.
Overall Survival (OS) | Up to approximately 2 years
  OS is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Wuhan Tongji Hospital, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi